CLINICAL TRIAL: NCT05539651
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of Subcutaneously Administered RBD5044 in Healthy Subjects
Brief Title: A Single and Multiple Ascending Doses Study to Evaluate the Safety and Pharmacokinetics of RBD5044
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Ribo Life Science Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBAP1101
Record Dates: First submitted 2022-08-22; First posted 2022-09-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Health Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RBD5044 SAD experimental group (Experimental): Subjects in SAD experimental groups will receive a single subcutaneous injection of RBD5044 on Day 1.
  Interventions: Drug: RBD5044
- RBD5044 MAD experimental group (Experimental): Subjects in MAD experimental groups will receive one subcutaneous injection of RBD5044 on Day 1 and another subcutaneous injection of RBD5044 on Day 29.
  Interventions: Drug: RBD5044
- Placebo SAD group (Placebo Comparator): Subjects in SAD placebo groups will receive a single subcutaneous injection of placebo on Day 1.
  Interventions: Drug: Placebo
- Placebo MAD group (Placebo Comparator): Subjects in MAD placebo groups will receive one subcutaneous injection of placebo on Day 1 and another subcutaneous injection of placebo on Day 29.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBD5044 — Subcutaneously Administered RBD5044 in Healthy Subjects
  Arms: RBD5044 MAD experimental group; RBD5044 SAD experimental group
Drug: Placebo — Subcutaneously Administered Placebo in Healthy Subjects
  Arms: Placebo MAD group; Placebo SAD group

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I study to evaluate the safety, tolerability, PK profiles and PD effect of single and multiple ascending doses of subcutaneously administered RBD5044 in healthy subjects. The study will be performed in 2 phases: single ascending dose (SAD) phase and multiple ascending doses (MAD) phase in healthy subjects. There are 6 cohorts in SAD phases, the dose levels are 5mg, 20mg, 60mg, 90mg, 120mg and 150mg. There are 3 cohorts in MAD phases, the dose levels are 60mg, 90mg and 120mg.The decision to escalate to subsequent dose levels will be made by the SRC based on the review of all available safety information, including AEs, ECGs, vital signs, and clinical laboratory test results in each cohort.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria are met:

1. Willing to comply with protocol required visit schedule and visit requirements and provide written informed consent.
2. Male and female subjects, aged 18 to 65 years (inclusive).
3. Body mass index between 18 and 32 kg/m2, inclusive.
4. Fasting TG ≥ 0.9 mmol/L (80 mg/dL) and ≤ 3.4 mmol/L (300 mg/dL) at screening.
5. Fasting LDL-C < 4.9 mmol/L (<190 mg/dL) at screening.
6. Healthy as determined by pre-study medical history, physical examination, clinical laboratory assessments, and 12-lead electrocardiogram (ECG).
7. Satisfy one of the following:

   * Females: must be non-pregnant and non-lactating; surgically sterile, post-menopausal, abstinent, or if engaged in sexual relations of child-bearing potential, the subject is using an acceptable contraceptive method (refer to Section 4.6.3) for four weeks before, during, and for at least 6 months after the last dose of study drug administration.
   * Males: must be surgically sterile, abstinent, or if engaged in sexual relations of child-bearing potential, the subject is utilizing an acceptable contraceptive method (refer to Section 4.6.3)) during and for at least 6 months after the last dose of study drug administration.
8. Non-smokers and non-nicotine users for at least 90 days before screening

Exclusion Criteria:

A subject meeting any of the following exclusion criteria will not be allowed to participate in this study:

1. Any uncontrolled or serious disease, or any medical or surgical condition, may interfere with participation in the clinical study and/or put the subject at significant risk (according to the investigator's judgment) if he/she participates in the clinical study.
2. History or presence of cardiovascular disease (including peripheral artery and cerebrovascular disease).
3. Systolic blood pressure (SBP) > 140 mmHg and/or diastolic blood pressure (DBP) > 90 mmHg after 10 minutes of supine rest, unless determined by the investigator to be not clinically relevant.
4. Diagnosis of diabetes mellitus.
5. Received any medication or nutraceutical to alter serum lipids within 30 days before screening.
6. Active serious mental illness or psychiatric disorder, including but not limited to schizophrenia, bipolar disorder, or severe depression, which require current pharmacological intervention.
7. Alanine aminotransferase (ALT) and/or total bilirubin are above the upper limit of normal reference range (ULN); no investigator discretion and repeat assessments are allowed.
8. Aspartate aminotransferase (AST), alkaline phosphatase (ALP), or gamma-glutamyl transferase (GGT) > 2 × ULN (no investigator discretion); or, if AST, ALP, or GGT > ULN, but ≤ 2 × ULN and considered clinically relevant by the investigator.
9. Used prescription drugs within 14 days or 7 half-lives (whichever is longer) before the first dose of study drug.
10. Used over-the-counter medication, excluding routine vitamins, within 7 days before the first dose of the study drug, unless determined by the investigator to be not clinically relevant, and unlikely to impact blood lipids level.
11. Received an investigational product within 30 days or 7 half-lives (whichever is longer) before the first dose of the study drug or are in the follow-up of another clinical study. If subjects used advanced therapy (ASO/siRNA/gene therapy/cell therapy), it should be judged by the investigator.
12. Hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), syphilis infection, or positive hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus antibody (HCVAb), HIV antibody (HIVAb), treponema pallidum antibody (TP-Ab) at screening.
13. Clinically significant illness within 7 days before the first dose of the study drug.
14. Consume more than 14 (female) or 21 (male) units of alcohol per week (unit: 1 glass of wine [125 mL] = 1 measure of spirits = ½ pint of beer) within the 12 months before screening or positive screen for alcohol abuse.
15. History or clinical evidence of drug abuse within the 12 months before screening or positive screen for drug abuse. Drug abuse is defined as compulsive, repetitive, and/or chronic use of drugs or other substances with or without problems related to their use and/or where stopping or a dose reduction will lead to withdrawal symptoms.
16. Donated more than 500 mL of blood within 90 days before the first dose of the study drug.
17. History of multiple drug allergies or history of allergic reaction to an oligonucleotide or N-acetylgalactosamine (GalNAc).
18. History of intolerance to subcutaneous (SC) injection or relevant abdominal scarring (surgical, burns, etc.).
19. Any conditions which would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | SAD: Up to 24 weeks; MAD: Up to 28 weeks
  The investigator will make an assessment of intensity for each AE and SAE reported during the study according to CTCAE V5.0

SECONDARY OUTCOMES:
To characterize the pharmacokinetic parameter Cmax of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  Plasma Maximum concentration (Cmax)
To characterize the pharmacokinetic parameter Tmax of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  Time to maximum concentration (Tmax)
To characterize the pharmacokinetic parameter AUC0-inf of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  Area under the concentration-time curve from 0 to infinity (inf) (AUC0-inf)
To characterize the pharmacokinetic parameter AUC0-t of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  Area under the concentration-time curve from 0 to the collection time t (AUC0-t)
To characterize the pharmacokinetic parameter t1/2 of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  Plasma Half-Life (t1/2)
To characterize the pharmacokinetic parameter λz of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  Terminal rate constant (λz)
To characterize the pharmacokinetic parameter MRT of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  mean residence time (MRT)
To characterize the pharmacokinetic parameter CL/F of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  Oral clearance (CL/F)
To characterize the pharmacokinetic parameter Vz/F of RBD5044 in healthy subjects | SAD: within 60 minutes before dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after dosing; MAD: within 60 minutes before day 1 and day 29 dosing, and at 0.25, 0.5, 1, 2, 4, 6, 8,10,12, 24 and 48 hours after Day 1 and day 29 dosing
  Volume of distribution in the terminal elimination period (Vz/F)
To evaluate the pharmacodynamics (PD) effect of RBD5044 on serum levels of APOC3 in healthy subjects | SAD: Up to 24 weeks; MAD: Up to 28 weeks
  by testing Concentrations of APOC3
To evaluate the PD effect of RBD5044 on serum levels of triglyceride (TG) in healthy subjects. | SAD: Up to 24 weeks; MAD: Up to 28 weeks
  by testing Concentrations of TG

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Limited, Brisbane, Australia